CLINICAL TRIAL: NCT05858112
Title: SuperTROPO (Better Diagnostics of Myocardial Infarction With a Test for Special Forms of Troponin)
Acronym: SuperTROPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Saara Wittfooth, Assistant professor, University of Turku
Other Study IDs: VARHA/487/13.02.02/2023
Record Dates: First submitted 2023-04-25; First posted 2023-05-15 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Infarction; Myocardial Ischemia
Keywords: Troponin; Myocardial ischemia; Myocardial infarction; High-sensitivity troponin T
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Leftover plasma from the blood samples collected routinely at the emergency department
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected MI
  Interventions: Diagnostic Test: SuperTROPO novel assay to measure the long forms of cTnT

INTERVENTIONS:
Diagnostic Test: SuperTROPO novel assay to measure the long forms of cTnT — SuperTROPO novel assay to measure the long forms of cTnT

SUMMARY:
The aim of this study is to investigate whether measurement of the long forms of cTnT with the novel SuperTROPO assay would improve the diagnosis of myocardial infarction in patients in the emergency department. The main goals are:

1. To assess whether measuring long forms of cTnT with the novel SuperTROPO assay and determining the ratio of long cTnT and standard high-sensitivity cTnT could separate patients with type 1 NSTEMI patients from patients with other causes of minor (> 14ng/L) cTnT elevation in a single admission blood sample in unselected emergency department patients with clinical indication for troponin measurement.
2. To compare the level of long cTnT and the ratio of long cTnT and standard cTnT in patients with type 1 MI and various clinical patient groups admitted to emergency department with elevated standard cTnT, e.g. patients with atrial fibrillation, heart failure or renal impairment.
3. To evaluate optimal cut-off values for long cTnT and its ratio to standard cTnT in the exclusion and diagnosis of MI in a clinical setting with elevated (>14ng/L) cTnT.
4. To evaluate how time from symptom onset and peak symptom to blood sampling, as well as comorbidities and patients' age impact the discriminative capacity of long cTnT and cTnT ratio between patients with and without type 1 MI.
5. To investigate whether information on long cTnT and its ratio to standard cTnT can be used to cut down unnecessary coronary angiographies and hospital admissions

The long forms of cTnT are measured from the residual blood samples routinely collected from patients with suspected myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patient has arrived at the emergency department and high-sensitivity cTnT test (P-TnT) has been ordered as part of the routine "cardiac package" of laboratory tests upon arrival
* Result of >14 ng/L of the P-TnT test included in the "cardiac package"
* Age > 18
* The patient or his/her legal representative has given written informed consent for participation in the study

Exclusion Criteria:

* unable to give informed consent
* legally incompetent individuals
* pregnancy
* previously participated in this study

Ages: 19 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department and suspected with myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarction type 1 | During the index hospitalization, that is, the hospitalization after the drawn blood samples at the emergency department. Up to 12 weeks.
  In brief, type 1 MI will be diagnosed when there is evidence of myocardial necrosis along with a clinical setting consistent with acute myocardial ischemia, as well as a coronary plaque rupture or erosion and superimposed thrombosis. The presence of the final diagnosis of type 1 MI by the treating clinician will be reviewed from patient records of the index hospitalization. Furthermore, patients with type 2 MI, will be identified and analyzed separately. The proportion of patients with type MI will be calculated and troponin values will be compared with patients with and without MI. .

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No